CLINICAL TRIAL: NCT01605916
Title: A Phase I, Open-Label Study to Investigate the Safety and Tolerability of AZD6244 (Selumetinib) When Given as a Monotherapy in Japanese Patients With Advanced Solid Malignancies, and When Given in Combination With Docetaxel as 2nd Line Therapy in Japanese Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (Stage IIIB-IV)
Brief Title: Investigate the Safety and Tolerability of AZD6244 Monotherapy or + Docetaxel in Japanese Patients With Advanced Solid Malignancies or Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1532C00067
Record Dates: First submitted 2012-05-21; First posted 2012-05-25 (Estimated); Results first posted 2016-07-14 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-09

CONDITIONS: Neoplasms,; Metastatic Cancer,; Non-Small Cell Lung Cancer; Advanced Solid Malignancies
Keywords: Cancer,; Tumour,; Metastatic,; Lung cancer,; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — AZD 6244

ARMS (5):
- Selumetinib (AZD6244) 25 mg (Experimental): monotherapy
  Interventions: Drug: AZD6244
- Selumetinib (AZD6244) 50 mg (Experimental): monotherapy
  Interventions: Drug: AZD6244
- Selumetinib (AZD6244) 75 mg (Experimental): monotherapy
  Interventions: Drug: AZD6244
- Selumetinib (AZD6244) 75 mg + Doce (Experimental): Combination
  Interventions: Drug: AZD6244
- Selumetinib (AZD6244) 25 mg + Doce (Experimental): combination
  Interventions: Drug: AZD6244

INTERVENTIONS:
Drug: AZD6244 — Tablet Oral bid
  Other Names: Selumetinib (AZD6244)

SUMMARY:
The objective of this study will be to investigate the safety and tolerability of AZD6244 given monotherapy or in combination with docetaxel as 2nd line therapy in Japanese patients with Advanced Solid Malignancies or Locally Advanced or Metastatic Non-Small Cell Lung Cancer. In addition, the pharmacokinetic profile of AZD6244 will be investigated. Following the combination regimen dose escalation phase (Part A) of the study additional patients may be enrolled to a dose expansion phase (Part B) to refine further the safety, tolerability, pharmacokinetics and biological activity of the combination in this patient population.

DETAILED DESCRIPTION:
The objective of the combination therapy part of this study will be to investigate the safety and tolerability of AZD6244 given in combination with docetaxel as 2nd line therapy in Japanese patients with Locally Advanced or Metastatic Non-Small Cell Lung Cancer (Stage IIIB-IV). In addition, the pharmacokinetic profile of AZD6244 and docetaxel will be investigated.

The objective of the monotherapy part of this study will be to investigate the safety and tolerability of AZD6244 given as a monotherapy in Japanese patients with advanced solid malignancies. In addition, the pharmacokinetic profile of monotherapy AZD6244 will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lung cancer who have not responded to prior therapy or have become worse.
* Patients who have overall good general conditions.
* Patients who have at least one lesion that can be accurately assessed by imaging.
* Patients who have appropriate renal conditions confirmed by test results for taking part in the study.
* Evidence of non-childbearing status for women of childbearing potential, or postmenopausal status.

Exclusion Criteria:

* Patients with brain metastases or spinal cord compression.
* Patients with significant abnormal ECG findings.
* Patients with evidence of severe or uncontrolled systemic disease.
* The main organ functional test values for bone marrow, kidney, and liver, etc., do not meet the standards.
* Patients with known hypersensitivity to docetaxel or products containing polysorbate 80.

Only for monotherapy cohort eligibility criteria Patients with advanced solid malignancies refractory to standard treatment or for which no standard therapy exists irrespective of the stage and previous treatment.

Patients with histologically or cytologically confirmed advanced solid malignancies.

Ages: 20 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-06; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Smith, Medical Science Director, Study Director — AstraZeneca; Yuichiro Ohe, Medical Doctor, Principal Investigator — National Cancer Centre East; Hideo Saka, Medical Doctor, Principal Investigator — National Hospital Organisation Nagoya Medical Centre; Takashi Seto, Medical Doctor, Principal Investigator — National Hospital Organization Kyushu Cancer Center
Locations (3):
- Japan (3):
  - Research Site, Fukuoka
  - Research Site, Kashiwa-shi
  - Research Site, Nagoya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled on 01 June 2012. Last subject last visit on 30 March 2015.
Pre-assignment Details: Out of 33 enrolled subjects, 25 subjects were assigned to selumetinib (AZD6244, ARRY-142886), and 8 subjects were not assigned. The reasons of no assignment were 'Screen failure' (7 subjects) and 'Withdrawal by subject' (1 subject).
Groups:
- Combination Therapy Cohort 1 Selumetinib 75 mg + Doce: Combination therapy of Selumetinib 75 mg twice a day with docetaxel 60 mg/m2 every 21 days for Japanese patients with locally advanced or metastatic non-small cell lung cancer
- Combination Therapy Cohort 2 Selumetinib 25 mg + Doce: Combination therapy of Selumetinib 25 mg twice a day with docetaxel 60 mg/m2 every 21 days for Japanese patients with locally advanced or metastatic non-small cell lung cancer
- Monotherapy Cohort 1 Selumetinib 25 mg: Monotherapy of Selumetinib 25 mg twice a day for Japanese patients with advanced solid malignancies
- Monotherapy Cohort 2 Selumetinib 50 mg: Monotherapy of Selumetinib 50 mg twice a day for Japanese patients with advanced solid malignancies
- Monotherapy Cohort 3 Selumetinib 75 mg: Monotherapy of Selumetinib 75 mg twice a day for Japanese patients with advanced solid malignancies
Period: Overall Study
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce | Monotherapy Cohort 1 Selumetinib 25 mg | Monotherapy Cohort 2 Selumetinib 50 mg | Monotherapy Cohort 3 Selumetinib 75 mg
Started | 4 | 4 | 4 | 6 | 7
Completed | 0 | 0 | 1 (Subject ongoing the study at data cut off) | 0 | 1 (Subject ongoing the study at data cut off)
Not Completed | 4 | 4 | 3 | 6 | 6
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 2 | 3 | 3 | 5 | 4
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All subjects who received selumetinib were included into the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce | Monotherapy Cohort 1 Selumetinib 25 mg | Monotherapy Cohort 2 Selumetinib 50 mg | Monotherapy Cohort 3 Selumetinib 75 mg | Total
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 7 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.5 (17.33) | 58.8 (8.50) | 60.0 (12.36) | 60.0 (11.75) | 66.7 (12.22) | 61.0 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 1 | 4 | 9
  Male | 3 | 3 | 2 | 5 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Selumetinib After Single Dose
Description: Pharmacokinetic parameter (Cmax: maximum plasma concentration) of Selumetinib following single oral dose of Selumetinib
Time Frame: Day 1: 0, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce | Monotherapy Cohort 1 Selumetinib 25 mg | Monotherapy Cohort 2 Selumetinib 50 mg | Monotherapy Cohort 3 Selumetinib 75 mg
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 7
ng/mL | 2534 (40.45) | 1073 (35.18) | 370.3 (96.87) | 897.1 (69.34) | 2084 (50.85)

2. Primary Outcome: Tmax of Selumetinib After Single Dose
Description: Pharmacokinetic parameter (tmax: time to reach the maximum plasma concentration) of Selumetinib following single oral dose of Selumetinib
Time Frame: Day 1: 0, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Median (Full Range); unit: hour
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce | Monotherapy Cohort 1 Selumetinib 25 mg | Monotherapy Cohort 2 Selumetinib 50 mg | Monotherapy Cohort 3 Selumetinib 75 mg
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 7
hour | 1.49 (40.45) [0.97 to 2.00] | 1.00 (35.18) [0.98 to 1.50] | 1.74 [0.47 to 4.05] | 1.51 [0.93 to 4.12] | 0.98 [0.93 to 2.00]

3. Primary Outcome: AUC(0-12) of Selumetinib After Single Dose
Description: Pharmacokinetic parameter (AUC(0-12): area under the plasma concentration-time curve from zero to 12 hours post-dosey) of Selumetinib following single oral dose of Selumetinib
Time Frame: Day 1: 0, 0.5, 1, 1.5, 2, 4, 8, 12 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce | Monotherapy Cohort 1 Selumetinib 25 mg | Monotherapy Cohort 2 Selumetinib 50 mg | Monotherapy Cohort 3 Selumetinib 75 mg
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 7
ng*h/mL | 6784 (26.63) | 1599 (35.48) | 1021 (30.62) | 2723 (33.24) | 5578 (35.77)

4. Primary Outcome: Cmax of N-desmethyl Selumetinib After Single Dose
Description: Pharmacokinetic parameter (Cmax: maximum plasma concentration) of N-desmethyl Selumetinib following single oral dose of Selumetinib
Time Frame: Day 1: 0, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce | Monotherapy Cohort 1 Selumetinib 25 mg | Monotherapy Cohort 2 Selumetinib 50 mg | Monotherapy Cohort 3 Selumetinib 75 mg
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 7
ng/mL | 130.8 (63.44) | 68.61 (15.10) | 27.50 (41.42) | 46.55 (57.74) | 136.6 (29.28)

5. Primary Outcome: Tmax of N-desmethyl Selumetinib After Single Dose
Description: Pharmacokinetic parameter (tmax: time to reach the maximum plasma concentration) of N-desmethyl Selumetinib following single oral dose of Selumetinib
Time Frame: Day 1: 0, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Median (Full Range); unit: hour
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce | Monotherapy Cohort 1 Selumetinib 25 mg | Monotherapy Cohort 2 Selumetinib 50 mg | Monotherapy Cohort 3 Selumetinib 75 mg
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 7
hour | 1.75 (40.45) [1.47 to 2.00] | 1.00 (35.18) [0.98 to 1.50] | 1.74 [0.47 to 4.05] | 1.75 [0.93 to 4.12] | 1.47 [0.93 to 2.00]

6. Primary Outcome: AUC(0-12) of N-desmethyl Selumetinib After Single Dose
Description: Pharmacokinetic parameter (AUC(0-12): area under the plasma concentration-time curve from zero to 12 hours post-dose) of N-desmethyl Selumetinib following single oral dose of Selumetinib
Time Frame: Day 1: 0, 0.5, 1, 1.5, 2, 4, 8, 12 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce | Monotherapy Cohort 1 Selumetinib 25 mg | Monotherapy Cohort 2 Selumetinib 50 mg | Monotherapy Cohort 3 Selumetinib 75 mg
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 7
ng*h/mL | 409.6 (32.29) | 159.6 (33.22) | 88.79 (7.700) | 182.6 (48.45) | 495.4 (17.99)

7. Primary Outcome: Cmax of Selumetinib During Oral Twice Daily Dose of Selumetinib
Description: Pharmacokinetic parameter (Cmax: maximum plasma concentration) of Selumetinib during oral twice daily dose of Selumetinib
Time Frame: Day 8: 0, 0.5, 1, 1.5, 2, 4, 8, 12 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce | Monotherapy Cohort 1 Selumetinib 25 mg | Monotherapy Cohort 2 Selumetinib 50 mg | Monotherapy Cohort 3 Selumetinib 75 mg
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 6
ng/mL | 2437 (64.93) | 662.3 (31.07) | 623.4 (46.09) | 1012 (47.08) | 2178 (79.67)

8. Primary Outcome: Tmax of Selumetinib During Oral Twice Daily Dose of Selumetinib
Description: Pharmacokinetic parameter (tmax: time to reach the maximum plasma concentration) of Selumetinib during oral twice daily dose of Selumetinib
Time Frame: Day 8: 0, 0.5, 1, 1.5, 2, 4, 8, 12 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Median (Full Range); unit: hour
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce | Monotherapy Cohort 1 Selumetinib 25 mg | Monotherapy Cohort 2 Selumetinib 50 mg | Monotherapy Cohort 3 Selumetinib 75 mg
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 6
hour | 3.97 (40.45) [1.48 to 4.02] | 1.25 (35.18) [1.00 to 12.00] | 1.23 [0.50 to 2.07] | 1.96 [1.00 to 4.03] | 1.50 [0.95 to 2.00]

9. Primary Outcome: AUC(0-12) of Selumetinib During Oral Twice Daily Dose of Selumetinib
Description: Pharmacokinetic parameter (AUC(0-12): area under the plasma concentration-time curve from zero to 12 hours post-dose) of Selumetinib during oral twice daily dose of Selumetinib
Time Frame: Day 8: 0, 0.5, 1, 1.5, 2, 4, 8, 12 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce | Monotherapy Cohort 1 Selumetinib 25 mg | Monotherapy Cohort 2 Selumetinib 50 mg | Monotherapy Cohort 3 Selumetinib 75 mg
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 6
ng*h/mL | 13050 (12.86) | 2334 (42.31) | 2130 (20.09) | 4818 (20.07) | 8734 (55.99)

10. Primary Outcome: Cmax of N-desmethyl Selumetinib During Oral Twice Daily Dose of Selumetinib
Description: Pharmacokinetic parameter (Cmax: maximum plasma concentration) of N-desmethyl Selumetinib during oral twice daily dose of Selumetinib
Time Frame: Day 8: 0, 0.5, 1, 1.5, 2, 4, 8, 12 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce | Monotherapy Cohort 1 Selumetinib 25 mg | Monotherapy Cohort 2 Selumetinib 50 mg | Monotherapy Cohort 3 Selumetinib 75 mg
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 6
ng/mL | 38.91 (133.7) | 34.46 (35.21) | 36.16 (31.26) | 42.18 (56.89) | 84.56 (74.73)

11. Primary Outcome: Tmax of N-desmethyl Selumetinib During Oral Twice Daily Dose of Selumetinib
Description: Pharmacokinetic parameter (tmax: time to reach the maximum plasma concentration) of N-desmethyl Selumetinib during oral twice daily dose of Selumetinib
Time Frame: Day 8: 0, 0.5, 1, 1.5, 2, 4, 8, 12 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Median (Full Range); unit: hour
Groups:
- Monotherapy Cohort 3 Selumetinib 75 mg: Monotherapy of Selumetinib 50 mg twice a day for Japanese patients with advanced solid malignancies
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce | Monotherapy Cohort 1 Selumetinib 25 mg | Monotherapy Cohort 2 Selumetinib 50 mg | Monotherapy Cohort 3 Selumetinib 75 mg
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 6
hour | 3.97 (40.45) [1.48 to 4.02] | 1.25 (35.18) [1.00 to 1.97] | 1.25 [0.95 to 2.07] | 1.96 [1.48 to 4.03] | 1.74 [0.98 to 4.00]

12. Primary Outcome: AUC(0-12) of N-desmethyl Selumetinib During Oral Twice Daily Dose of Selumetinib
Description: Pharmacokinetic parameter (AUC(0-12): area under the plasma concentration-time curve from zero to 12 hours post-dose) of N-desmethyl Selumetinib during oral twice daily dose of Selumetinib
Time Frame: Day 8: 0, 0.5, 1, 1.5, 2, 4, 8, 12 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce | Monotherapy Cohort 1 Selumetinib 25 mg | Monotherapy Cohort 2 Selumetinib 50 mg | Monotherapy Cohort 3 Selumetinib 75 mg
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 6
ng*h/mL | 241.5 (115.7) | 150.4 (44.08) | 146.3 (29.77) | 251.3 (39.33) | 445.0 (61.88)

13. Secondary Outcome: Cmax of Docetaxel Following Intravenous Infusion of Docetaxel 60 mg/m2
Description: Pharmacokinetic parameter (Cmax: maximum plasma concentration) of docetaxel following intravenous infusion of docetaxel 60 mg/m2 in combination with Selumetinib
Time Frame: Day 1: 0, 0.5, 1, 1.5, 2, 4, 8, 12 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce
Number analyzed (Participants) | 4 | 4
ng/mL | 2329 (9.805) | 2726 (27.92)

14. Secondary Outcome: Tmax of Docetaxel Following Intravenous Infusion of Docetaxel 60 mg/m2
Description: Pharmacokinetic parameter (tmax: time to reach the maximum plasma concentration) of docetaxel following intravenous infusion of docetaxel 60 mg/m2 in combination with Selumetinib
Time Frame: Day 1: 0, 0.5, 1, 1.5, 2, 4, 8, 12 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Median (Full Range); unit: hour
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce
Number analyzed (Participants) | 4 | 4
hour | 0.99 (9.805) [0.50 to 1.05] | 0.99 (27.92) [0.93 to 1.00]

15. Secondary Outcome: AUC(0-12) of Docetaxel Following Intravenous Infusion of Docetaxel 60 mg/m2
Description: Pharmacokinetic parameter (AUC(0-12): area under the plasma concentration-time curve from zero to 12 hours post-dose) of docetaxel following intravenous infusion of docetaxel 60 mg/m2 in combination with Selumetinib
Time Frame: Day 1: 0, 0.5, 1, 1.5, 2, 4, 8, 12 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce
Number analyzed (Participants) | 4 | 4
ng*h/mL | 2422 (13.72) | 3056 (28.64)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study, from informed consent until the end of the followup period. The follow-up period is defined as 28 days after investigational prooduct and/or docetaxel is discontinued.
Arm/Group | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce | Monotherapy Cohort 1 Selumetinib 25 mg | Monotherapy Cohort 2 Selumetinib 50 mg | Monotherapy Cohort 3 Selumetinib 75 mg
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 1/4 | 1/6 | 2/7
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce (N=4) | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce (N=4) | Monotherapy Cohort 1 Selumetinib 25 mg (N=4) | Monotherapy Cohort 2 Selumetinib 50 mg (N=6) | Monotherapy Cohort 3 Selumetinib 75 mg (N=7)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy Cohort 1 Selumetinib 75 mg + Doce (N=4) | Combination Therapy Cohort 2 Selumetinib 25 mg + Doce (N=4) | Monotherapy Cohort 1 Selumetinib 25 mg (N=4) | Monotherapy Cohort 2 Selumetinib 50 mg (N=6) | Monotherapy Cohort 3 Selumetinib 75 mg (N=7)
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nail infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 1 | 0
Food allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Delusion (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 2
Eye oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 2 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 1 | 0
Xanthopsia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Vascular pain (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 1 | 2 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 0 | 2 | 2
Stomatitis (Gastrointestinal disorders) | 4 | 1 | 0 | 1 | 2
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 1 | 4 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 3 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 2
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 2
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 2 | 1 | 3 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 1 | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 3
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 1 | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 1 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 3 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 2 | 3 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs were prohibited to disclose all information related to this study without AZ approval before this study was completed.